CLINICAL TRIAL: NCT01431794
Title: Phase 1/2 Safety and Feasibility of Gemcitabine and Nab-Paclitaxel in Combination With LDE-225 as Neoadjuvant Therapy in Patients With Borderline Resectable Pancreatic Adenocarcinoma.
Brief Title: Gemcitabine + Nab-paclitaxel With LDE-225 (Hedgehog Inhibitor) as Neoadjuvant Therapy for Pancreatic Adenocarcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to cease in manufacturing of study drug.
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Novartis Pharmaceuticals (Industry); The Skip Viragh Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1130; NA_00047491 (Other: JHMIRB)
Record Dates: First submitted 2011-07-19; First posted 2011-09-12 (Estimated); Results first posted 2019-06-25 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Pancreatic Ductal Adenocarcinoma
Keywords: Pancreatic ductal adenocarcinoma (PDA)Neoplasms; LDE225; nab-paclitaxel; abraxane; gemcitabine; neoadjuvant; cytotoxic; hedgehog inhibitor; stromal cells; resectable PDA; Pancreatic Diseases; Carcinoma; Sonidegib
MeSH Terms: conditions — Pancreatic Diseases; Carcinoma | interventions — sonidegib; Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase I-Gem,nab-paclitaxel,LDE225-600mg (Experimental): Four cycles of Gemcitabine (gem) 1000 mg/m2 and nab-Paclitaxel 125 mg/ m2 on days 1, 8, and 15 every 28 days cycle in combination with escalating doses of oral LDE225 (Sonidegib), 600 mg daily.
  Interventions: Drug: LDE225-600mg; Drug: Gemcitabine; Drug: nab-paclitaxel
- Phase II-Arm A:Gem,nab-paclitaxel,LDE225 (Active Comparator): Four cycles of gemcitabine 1000 mg/m2 and nab-Paclitaxel 125 mg/m2 on days 1, 8 and 15 in combination with LDE-225 at the recommended phase 2 dose. Cycles repeated every 28 days.
  Interventions: Drug: LDE225-600mg; Drug: Gemcitabine; Drug: nab-paclitaxel; Drug: LDE225-400mg; Drug: LDE225-800mg
- Phase II-Arm B:Gem,nab-paclitaxel (Active Comparator): Four cycles of gemcitabine 1000 mg/m2 and nab-Paclitaxel 125 mg/m2 on days 1, 8 and 15. Cycles repeated every 28 days.
  Interventions: Drug: Gemcitabine; Drug: nab-paclitaxel
- Phase I-Gem,nab-paclitaxel,LDE225-400mg (Experimental): Four cycles of Gemcitabine (gem) 1000 mg/m2 and nab-Paclitaxel 125 mg/ m2 on days 1, 8, and 15 every 28 days cycle in combination with escalating doses of oral LDE225 (Sonidegib), 400 mg daily.
  Interventions: Drug: Gemcitabine; Drug: nab-paclitaxel; Drug: LDE225-400mg
- Phase I-Gem,nab-paclitaxel,LDE225-800mg (Experimental): Four cycles of Gemcitabine (gem) 1000 mg/m2 and nab-Paclitaxel 125 mg/ m2 on days 1, 8, and 15 every 28 days cycle in combination with escalating doses of oral LDE225 (Sonidegib), 800 mg daily.
  Interventions: Drug: Gemcitabine; Drug: nab-paclitaxel; Drug: LDE225-800mg

INTERVENTIONS:
Drug: LDE225-600mg — Phase I: oral LDE225 (Sonidegib), 600mg daily.
  Phase II Arm A: LDE225 at the recommended phase 2 dose on Days 1, 8 and 15. Cycles repeated every 28 days.
  Other Names: Sonidegib
  Arms: Phase I-Gem,nab-paclitaxel,LDE225-600mg; Phase II-Arm A:Gem,nab-paclitaxel,LDE225
Drug: Gemcitabine — Four cycles of Gemcitabine 1000 mg/m2 on days 1, 8, and 15 every 28 days.
  Other Names: gem
Drug: nab-paclitaxel — Four cycles of nab-Paclitaxel 125 mg/m2 on days 1, 8, and 15 every 28 days.
  Other Names: abraxane
Drug: LDE225-400mg — Phase I: oral LDE225 (Sonidegib), 400mg daily.
  Other Names: Sonidegib
  Arms: Phase I-Gem,nab-paclitaxel,LDE225-400mg; Phase II-Arm A:Gem,nab-paclitaxel,LDE225
Drug: LDE225-800mg — Phase I: oral LDE225 (Sonidegib), 800mg daily.
  Other Names: Sonidegib
  Arms: Phase I-Gem,nab-paclitaxel,LDE225-800mg; Phase II-Arm A:Gem,nab-paclitaxel,LDE225

SUMMARY:
This is an open-label phase 1/2 study that will combine the chemotherapy agents gemcitabine and nab-paclitaxel with an oral hedgehog inhibitor LDE225 (Sonidegib). The objective is to assess tolerability and the resection rate of patients with borderline resectable pancreatic adenocarcinoma who use this treatment.

DETAILED DESCRIPTION:
The investigators propose treating 6-12 patients during the phase 1 portion and 40 patients in the phase 2 stage.

Phase 1 Stage:

Four cycles of gemcitabine 1000 mg/m2 and nab-paclitaxel 125 mg/m2 on days 1, 8 and 15 in combination with escalating doses (400mg, or 600mg, or 800mg) of LDE-225. After completion of neoadjuvant therapy, the subjects will receive combined chemotherapy and radiation. Then subjects who are eligible for resection will go ahead with surgery. Following resection, subjects will complete two additional cycles of gemcitabine 1000 mg/m2 and nab-paclitaxel 125 mg/m2 in combination with LDE-225.

Phase 2 Stage: In the Phase 2 stage the patients will be randomized to receive gemcitabine and nab-paclitaxel with or without the hedgehog inhibitor LDE225:

1. Arm A: Four cycles of gemcitabine 1000 mg/m2 and nab-paclitaxel 125 mg/m on days 1, 8 and 15 in combination with LDE-225 at the recommended phase 2 dose.
2. Arm B: Four cycles of gemcitabine 1000 mg/m2 and nab-paclitaxel 125 mg/m on days 1, 8 and 15.

After completion of neoadjuvant therapy, the subjects will receive combined chemotherapy and radiation. Then subjects who are eligible for resection will go ahead with surgery. Following resection, subjects will complete two additional cycles of the pre-surgical therapy.

Several correlative laboratory studies will be conducted during the course of this study. They were designed around the goals of providing us with a better understanding of how the stroma-tumor interaction and the intra-tumoral drug levels of gemcitabine are affected with the use of LDE-225. Two additional biopsies are required to participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the pancreas.
* Must have borderline resectable pancreatic adenocarcinoma
* Measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension
* No previous radiotherapy, surgery, chemotherapy or investigational drug therapy.
* Age >18 years
* Life expectancy of greater than 1 month.
* ECOG (Eastern Cooperative Oncology Group) performance status 0 or 1
* Adequate organ and marrow function
* Asymptomatic for jaundice and ascites. Pain symptoms should be stable.
* Negative serum pregnancy test
* Sexually active males should agree to use a barrier form of contraception, even if they have had a vasectomy, during the study and for 6 months after stopping LDE225. Males should not donate sperm during treatment, and for up to six months after last dose. Sexually active females of child bearing potential agree to using highly effective contraception during study and for 20 months after final dose of LDE225.
* Agree not to donate blood products for 12 months after stopping LDE225.
* Willing to have two biopsies while on treatment for correlative studies.

Exclusion Criteria:

* Patients who have had previous radiotherapy, surgical resection, chemotherapy or investigational drug therapy for pancreatic adenocarcinoma.
* Patient has known metastatic disease.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to LDE225 or other agents used in the study.
* Patients taking medications with narrow therapeutic indices that are metabolized by cytochrome P450 (CYP450), including warfarin sodium (Coumadin®)
* Uncontrolled illness including, but not limited to, ongoing or active infection requiring IV antibiotics, symptomatic congestive heart failure not controlled with medication, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded
* Patient has undergone a major surgery, other than diagnostic surgery within four weeks prior to starting treatment on this study.
* Patients who are receiving treatment with medications known to be moderate and strong inhibitors or inducers of CYP3A4/5 or drugs metabolized by CYP2B6 or CYP2C9 that have narrow therapeutic index, and that cannot be discontinued before starting treatment with LDE225. Medications that are strong CYP3A4/5 inhibitors should be discontinued at least 7 days and strong CYP3A/5 inducers for at least 2 weeks prior to starting treatment with LDE225.
* Patients with neuromuscular disorders.
* Patients with impaired cardiac function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-12-27 (Actual); Primary Completion 2018-11-05 (Actual); Study Completion 2018-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana De Jesus-Acosta, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center JHMI
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10 subjects were screen failures. All of 13 subjects were enrolled into the Arm/group: Phase I: gem, nab-paclitaxel, and LDE225-600mg. Other Arm/group did not enroll any subjects due to early termination of the study.
Groups:
- Phase I: Gem, Nab-paclitaxel, and LDE225-600mg: Four cycles of Gemcitabine 1000 mg/m2 and nab-Paclitaxel 125 mg/m2 on days 1, 8, and 15 every 28 days cycle in combination with escalating doses of oral LDE225 (Sonidegib), 600 mg daily.
- Phase I: Gem, Nab-paclitaxel, and LDE225-400mg: Four cycles of Gemcitabine 1000 mg/m2 and nab-Paclitaxel 125 mg/m2 on days 1, 8, and 15 every 28 days cycle in combination with escalating doses of oral LDE225 (Sonidegib), 400 mg daily.
- Phase I: Gem, Nab-paclitaxel, and LDE225-800mg: Four cycles of Gemcitabine 1000 mg/m2 and nab-Paclitaxel 125 mg/m2 on days 1, 8, and 15 every 28 days cycle in combination with escalating doses of oral LDE225 (Sonidegib), 800 mg daily.
- Phase II: Arm A - Gem, Nab-paclitaxel, and LDE 225: Four cycles of gemcitabine 1000 mg/m2 and nab-Paclitaxel 125 mg/m2 on days 1, 8 and 15 in combination with LDE-225 at the recommended phase 2 dose. Cycles repeated every 28 days.
- Phase II: Arm B - Gemcitabine and Nab-paclitaxel: Four cycles of gemcitabine 1000 mg/m2 and nab-Paclitaxel 125 mg/m2 on days 1, 8 and 15. Cycles repeated every 28 days.
Period: Overall Study
Arm/Group | Phase I: Gem, Nab-paclitaxel, and LDE225-600mg | Phase I: Gem, Nab-paclitaxel, and LDE225-400mg | Phase I: Gem, Nab-paclitaxel, and LDE225-800mg | Phase II: Arm A - Gem, Nab-paclitaxel, and LDE 225 | Phase II: Arm B - Gemcitabine and Nab-paclitaxel
Started | 13 | 0 (not started due to early study's termination) | 0 (not started due to early study's termination) | 0 (not started due to early study's termination) | 0 (not started due to early study's termination)
Completed | 13 | 0 (not started due to early study's termination) | 0 (not started due to early study's termination) | 0 (not started due to early study's termination) | 0 (not started due to early study's termination)
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants were enrolled in Phase 1, gem, nab-paclitaxel, and LDE225-600mg arm only. Other arms did not have any participants due to the study's early termination.
Groups:
- Phase I, Gem, Nab-paclitaxel, and LDE225-600mg: Phase I:
  Four cycles of Gemcitabine 1000 mg/m2 and nab-Paclitaxel 125 mg/ m2 on days 1, 8, and 15 every 28 days cycle in combination with oral LDE225 600 mg daily
- Phase I, Gem, Nab-paclitaxel, and LDE225-400mg: Phase I:
  Four cycles of Gemcitabine 1000 mg/m2 and nab-Paclitaxel 125 mg/ m2 on days 1, 8, and 15 every 28 days cycle in combination with oral LDE225 400 mg daily
- Phase I, Gem, Nab-paclitaxel, and LDE225-800mg: Phase I:
  Four cycles of Gemcitabine 1000 mg/m2 and nab-Paclitaxel 125 mg/ m2 on days 1, 8, and 15 every 28 days cycle in combination with oral LDE225 800 mg daily
- Phase II, Arm A: Gem, Nab-paclitaxel, and LDE 225: Phase II:
  Arm A: Four cycles of gemcitabine 1000 mg/m2 and nab-Paclitaxel 125 mg/m2 on days 1, 8 and 15 in combination with LDE-225 at the recommended phase 2 dose from Phase I. Cycles repeated every 28 days.
- Phase II, Arm B: Gemcitabine and Nab-paclitaxel: Phase II:
  Arm B: Four cycles of gemcitabine 1000 mg/m2 and nab-Paclitaxel 125 mg/m2 on days 1, 8 and 15. Cycles repeated every 28 days.
- Total: Total of all reporting groups
Arm/Group | Phase I, Gem, Nab-paclitaxel, and LDE225-600mg | Phase I, Gem, Nab-paclitaxel, and LDE225-400mg | Phase I, Gem, Nab-paclitaxel, and LDE225-800mg | Phase II, Arm A: Gem, Nab-paclitaxel, and LDE 225 | Phase II, Arm B: Gemcitabine and Nab-paclitaxel | Total
Number analyzed (Participants) | 13 | 0 | 0 | 0 | 0 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.62 (9.32) |  |  |  |  | 61.62 (9.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 |  |  |  |  | 7
  Male | 6 |  |  |  |  | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino: White or Caucasian | 11 |  |  |  |  | 11
  Not Hispanic or Latino: Black or African American | 2 |  |  |  |  | 2
  Not Hispanic or Latino: Others | 0 |  |  |  |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Phase I - Safety and Feasibility of Gemcitabine and Nab-Paclitaxel in Combination With LDE-225 as Neoadjuvant Therapy as Measured by Number of Participants Who Tolerated the Maximal Dose of LDE-225
Description: Number of participants who tolerated the maximal dose of LDE-225 in combination with gemcitabine, nab-paclitaxel as neoadjuvant therapy in patients with borderline resectable pancreatic adenocarcinoma (PDA).
Time Frame: 5 years
Population: This measure only applies to the Phase I arms. All 13 subjects participated in the Arm/group: Phase I: gem, nab-paclitaxel, and LDE225-600mg. There were no participants enrolled in other two Arm/group as the study was terminated.
Measure: Count of Participants; unit: Participants
Groups:
- Phase I: Gem, Nab-paclitaxel, and LDE225-600mg: Four cycles of Gemcitabine (gem) 1000 mg/m2 and nab-Paclitaxel 125 mg/m2 on days 1, 8, and 15 every 28 days cycle in combination with escalating doses of oral LDE225 (Sonidegib), 600 mg daily.
- Phase I: Gem, Nab-paclitaxel, and LDE225-400mg: Four cycles of Gemcitabine (gem) 1000 mg/m2 and nab-Paclitaxel 125 mg/m2 on days 1, 8, and 15 every 28 days cycle in combination with escalating doses of oral LDE225 (Sonidegib), 400 mg daily.
- Phase I: Gem, Nab-paclitaxel, and LDE225-800mg: Four cycles of Gemcitabine (gem) 1000 mg/m2 and nab-Paclitaxel 125 mg/m2 on days 1, 8, and 15 every 28 days cycle in combination with escalating doses of oral LDE225 (Sonidegib), 800 mg daily.
Arm/Group | Phase I: Gem, Nab-paclitaxel, and LDE225-600mg | Phase I: Gem, Nab-paclitaxel, and LDE225-400mg | Phase I: Gem, Nab-paclitaxel, and LDE225-800mg
Number analyzed (Participants) | 13 | 0 | 0
Participants | 13 | 0 | 0

2. Primary Outcome: Phase II - Resection Rate of Two Preoperative Chemotherapy Regimens in Patients With Borderline Resectable PDA
Description: Number of participants with borderline resectable pancreatic adenocarcinoma (PDA) who undergo resection after therapy
Time Frame: 5 years
Population: No data was collected to assess this outcome measure as the study was terminated before Phase II.
Groups:
- Phase II-Arm A:Gem,Nab-paclitaxel,LDE225: Four cycles of gemcitabine 1000 mg/m2 and nab-Paclitaxel 125 mg/m2 on days 1, 8 and 15 in combination with LDE-225 at the recommended phase 2 dose. Cycles repeated every 28 days.
  LDE225-600mg: Phase I: oral LDE225 (Sonidegib), 600mg daily.
  Phase II Arm A: LDE225 at the recommended phase 2 dose on Days 1, 8 and 15. Cycles repeated every 28 days.
  Gemcitabine: Four cycles of Gemcitabine 1000 mg/m2 on days 1, 8, and 15 every 28 days.
  nab-paclitaxel: Four cycles of nab-Paclitaxel 125 mg/m2 on days 1, 8, and 15 every 28 days.
  LDE225-400mg: Phase I: oral LDE225 (Sonidegib), 400mg daily.
  LDE225-800mg: Phase I: oral LDE225 (Sonidegib), 800mg daily.
Arm/Group | Phase II-Arm A:Gem,Nab-paclitaxel,LDE225 | Phase II-Arm B:Gem,Nab-paclitaxel
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Overall Survival
Description: Number of months alive from cycle 1, Day 1 until 5 years post-intervention or death, whichever comes first.
Time Frame: 5 years
Population: as for outcome 1
Measure: Median (Full Range); unit: months
Arm/Group | Phase I: Gem, Nab-paclitaxel, and LDE225-600mg | Phase I: Gem, Nab-paclitaxel, and LDE225-400mg | Phase I: Gem, Nab-paclitaxel, and LDE225-800mg
Number analyzed (Participants) | 13 | 0 | 0
months | 34.3 [3.7 to 60] |  |

4. Secondary Outcome: Overall Tumor Response as Determined by Number of Participants With Complete or Partial Response
Description: Number of participants who experienced complete response (CR) or partial response (PR), as defined by RECIST v1.0; where CR is a disappearance of all target lesions and PR is ≥30% reduction of target lesions.
Time Frame: 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: Gem, Nab-paclitaxel, and LDE225-600mg | Phase I: Gem, Nab-paclitaxel, and LDE225-400mg | Phase I: Gem, Nab-paclitaxel, and LDE225-800mg
Number analyzed (Participants) | 13 | 0 | 0
Participants | 3 |  |

ADVERSE EVENTS:
Time Frame: up to 3 years
Description: Only for eligible participants. There were no participants enrolled in Phase I: gem, nab-paclitaxel, and LDE225-400mg, Phase I: gem, nab-paclitaxel, and LDE225-800mg, Phase II Arm A, and Phase II Arm B because the study was terminated early
Groups:
- Phase I, Gem, Nab-paclitaxel, and LDE225-600mg: Four cycles of Gemcitabine 1000 mg/m2 and nab-Paclitaxel 125 mg/ m2 on days 1, 8, and 15 every 28 days cycle with oral LDE225, 600mg.
- Phase I, Gem, Nab-paclitaxel, and LDE225-400mg: Four cycles of Gemcitabine 1000 mg/m2 and nab-Paclitaxel 125 mg/ m2 on days 1, 8, and 15 every 28 days cycle with oral LDE225, 400mg.
- Phase I, Gem, Nab-paclitaxel, and LDE225-800mg: Four cycles of Gemcitabine 1000 mg/m2 and nab-Paclitaxel 125 mg/ m2o n days 1, 8, and 15 every 28 days cycle with oral LDE225, 800mg.
- Phase II, Arm A: Gem, Nab-paclitaxel, and LDE 225: Phase II:
  Arm A: Four cycles of gemcitabine 1000 mg/m2 and nab-Paclitaxel 125 mg/m2 on days 1, 8 and 15 in combination with LDE-225 at the recommended phase I dose. Cycles repeated every 28 days.
Arm/Group | Phase I, Gem, Nab-paclitaxel, and LDE225-600mg | Phase I, Gem, Nab-paclitaxel, and LDE225-400mg | Phase I, Gem, Nab-paclitaxel, and LDE225-800mg | Phase II, Arm A: Gem, Nab-paclitaxel, and LDE 225 | Phase II, Arm B: Gemcitabine and Nab-paclitaxel
All-Cause Mortality (participants affected / at risk) | 2/13 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 8/13 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 13/13 | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I, Gem, Nab-paclitaxel, and LDE225-600mg (N=13) | Phase I, Gem, Nab-paclitaxel, and LDE225-400mg (N=0) | Phase I, Gem, Nab-paclitaxel, and LDE225-800mg (N=0) | Phase II, Arm A: Gem, Nab-paclitaxel, and LDE 225 (N=0) | Phase II, Arm B: Gemcitabine and Nab-paclitaxel (N=0)
nausea, vomitting (General disorders) | 3 (3) | NA | NA | NA | NA
abdomina pain (Gastrointestinal disorders) | 3 (3) | NA | NA | NA | NA
rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | NA | NA | NA | NA
fever and tachydysrhythmia (Cardiac disorders) | 1 (1) | NA | NA | NA | NA
spesis (Infections and infestations) | 1 (1) | NA | NA | NA | NA
obstruction (Gastrointestinal disorders) | 1 (1) | NA | NA | NA | NA
toxic mega-colon (Gastrointestinal disorders) | 1 (1) | NA | NA | NA | NA
pancreatitis (Gastrointestinal disorders) | 1 (1) | NA | NA | NA | NA
elevated creatine kinase (Blood and lymphatic system disorders) | 1 (1) | NA | NA | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I, Gem, Nab-paclitaxel, and LDE225-600mg (N=13) | Phase I, Gem, Nab-paclitaxel, and LDE225-400mg (N=0) | Phase I, Gem, Nab-paclitaxel, and LDE225-800mg (N=0) | Phase II, Arm A: Gem, Nab-paclitaxel, and LDE 225 (N=0) | Phase II, Arm B: Gemcitabine and Nab-paclitaxel (N=0)
WBC decreased (Blood and lymphatic system disorders) | 13 (68) | NA | NA | NA | NA — count of white blood cells
Hemoglobin decreased (Blood and lymphatic system disorders) | 12 (60) | NA | NA | NA | NA — hemoglobin count decreased and anemia
ALT increased (Hepatobiliary disorders) | 12 (30) | NA | NA | NA | NA — alanine aminotransferase level increased
sodium decreased (Metabolism and nutrition disorders) | 9 (9) | NA | NA | NA | NA — sodium ion decreased
Glucose increased (Metabolism and nutrition disorders) | 12 (52) | NA | NA | NA | NA — blood glucose level increased
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 10 (28) | NA | NA | NA | NA — alkaline phosphatase level increased
Albumin decreased (Blood and lymphatic system disorders) | 8 (23) | NA | NA | NA | NA
AST increased (Hepatobiliary disorders) | 10 (34) | NA | NA | NA | NA — Aspartate aminotransferase level increased
Calcium decreased (Metabolism and nutrition disorders) | 10 (20) | NA | NA | NA | NA — calcium ion in blood decreased
Lymphocytes decreased (Blood and lymphatic system disorders) | 10 (51) | NA | NA | NA | NA
Neutrophiles decreased (Blood and lymphatic system disorders) | 10 (32) | NA | NA | NA | NA
Platelets decreased (Blood and lymphatic system disorders) | 8 (23) | NA | NA | NA | NA — platelets count decreased
Anorexia (Metabolism and nutrition disorders) | 10 (28) | NA | NA | NA | NA
Weight loss (General disorders) | 10 (19) | NA | NA | NA | NA
Nausea (General disorders) | 10 (23) | NA | NA | NA | NA
Fatigue (General disorders) | 9 (24) | NA | NA | NA | NA
Constipation (Gastrointestinal disorders) | 8 (15) | NA | NA | NA | NA
Abdomin pain (Gastrointestinal disorders) | 7 (21) | NA | NA | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 7 (8) | NA | NA | NA | NA
Fever (General disorders) | 7 (10) | NA | NA | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-08-13): https://cdn.clinicaltrials.gov/large-docs/94/NCT01431794/Prot_SAP_000.pdf